CLINICAL TRIAL: NCT01099605
Title: Continuous Infusion of Local Anesthetic for Optimal Post Operative Pain Control Following Hemorrhoidectomy: A Randomized Double-blind Controlled Trial
Brief Title: Continuous Infusion of Local Anesthetic for Optimal Post Operative Pain Control Following Hemorrhoidectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No recruitment occurred and PI stopped the study
Sponsor: United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP# 10.0042
Record Dates: First submitted 2010-04-06; First posted 2010-04-07 (Estimated); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Hemorrhoids
Keywords: hemorrhoidectomy; pain management
MeSH Terms: conditions — Hemorrhoids; Agnosia

STUDY DESIGN:
Intervention Model Description: Bupivacaine vs pump
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pump device (Placebo Comparator): One arm will have continuous subcutaneous infusion of normal saline.
  Interventions: Device: placement of a continuous infusion pump
- Bupivacaine (Active Comparator): will receive continuous infusion of bupivacaine
  Interventions: Device: continuous infusion pump of bupivacaine

INTERVENTIONS:
Device: placement of a continuous infusion pump — Each infusion pump is placed below the mucosa of the rectum. Infusion of either the drug or saline will continue for approximately 3-4 days.
  Arms: Pump device
Device: continuous infusion pump of bupivacaine — bupivacaine 0.25% at 4ml/hr for 3 to 4 days
  Arms: Bupivacaine

SUMMARY:
Over the past decade, continuous wound infiltration systems have been introduced to treat a variety of post-surgical pain. These systems, commonly referred to pain pumps by patients, possess a catheter(s) attached to a reservoir of local anesthetic that directly infuses into the surgical site to provide local pain control thus avoiding the common and less desirable systemic effects of oral narcotic pain medication. Due to its portability, another benefit associated with these wound infiltration systems is its use as an outpatient pain control modality. Despite the apparent benefits, the verdict on the system's effectiveness in treating pain - throughout a variety of surgical fields - varies between very effective in reducing post-operative pain and reducing overall narcotic consumption for several days to completely ineffective with no reported changes in perceived pain or overall narcotic use.

Through a randomized trial comparing plain saline to a common local anesthetic, The investigators hope to evaluate the effectiveness of these pain pumps as an outpatient modality for pain management following hemorrhoidectomy patients. The investigators hypothesize that there will be a significant benefit in pain relief with the use of these pumps.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for hemorrhoidectomies at NMCP

Exclusion Criteria:

* Any patient with co-existing active purulent infection (i.e. abscess).
* Any patient who has had previous surgical intervention for his/her hemorrhoidal disease. Previous simple incision to treat a thrombosed hemorrhoid is not considered a surgical intervention for the purposes of this study. The minimal scar produced by a small incision would not alter post-operative pain following removal of a hemorrhoidal column.
* Any patient allergic to local anesthetics or oral pain medications
* Any patient with a history of chronic pain
* Any patient allergic to or has had an adverse reaction (i.e. history of gastrointestinal bleed) to a non-steroidal anti-inflammatory drugs (NSAIDs)
* Any patient pregnant patient

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03-10 (Actual); Primary Completion 2013-09-09 (Actual); Study Completion 2013-09-09 (Actual)

PRIMARY OUTCOMES:
VAS pain scales | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Medical Center Portsmouth, Portsmouth, Virginia, United States